CLINICAL TRIAL: NCT06790875
Title: Effects of Low Tidal Volume and Airway Pressure Release Ventilation on Lung Tissue Mechanics in ARDS Patients Under Mechanical Ventilation: A Prospective Randomized Crossover Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, XiaoJing Zou,MD, Principal Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EITDRRS
Record Dates: First submitted 2025-01-10; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome)
Keywords: ARDS; MP; DRRS
MeSH Terms: conditions — Acute Lung Injury | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Airway Pressure Release Ventilation (APRV)
  Interventions: Device: Airway Pressure Release Ventilation (APRV)
- Control group (No Intervention): Low tidal volume ventilation

INTERVENTIONS:
Device: Airway Pressure Release Ventilation (APRV) — In this arm, participants will receive airway pressure release ventilation (APRV), a form of pressure-controlled mechanical ventilation. The high pressure (Phigh) is set based on the plateau pressure of the LTV mode, with a low pressure (Plow) set at 0 cmH₂O. The high pressure time (Thigh) will be set to 4-6 seconds to maintain alveolar recruitment, while the low pressure time (Tlow) will be set to 0.2-0.6 seconds to optimize expiratory flow. This arm aims to evaluate the effects of APRV on lung tissue mechanics, oxygenation, and overall respiratory function in ARDS patients.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn how low tidal volume ventilation (LTV) and airway pressure release ventilation (APRV) affect lung tissue mechanics in adults with ARDS. The main questions it aims to answer are:

Does LTV or APRV improve lung tissue mechanics in patients with ARDS under mechanical ventilation? Researchers will compare LTV and APRV to see which ventilation mode works better for improving lung mechanics and patient safety.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria of the 2023 Global New Definition of ARDS.
2. Age: 18-80 years.
3. PaO2/FiO2 ≤ 200.
4. Within 12 hours of invasive mechanical ventilation treatment.
5. Obtain consent from the patient or their family members to participate in the study, and sign the informed consent form.

Exclusion Criteria:

1. Age < 18 years or > 80 years.
2. Uncorrected shock of any type.
3. Chronic obstructive pulmonary disease (COPD), pulmonary embolism, right heart failure, pulmonary hypertension, or severe arrhythmia.
4. Contraindications for using Electrical Impedance Tomography (EIT) (extensive chest skin damage, infection, pacemaker implantation, implanted automatic defibrillator, etc.), pneumothorax, mediastinal emphysema, or large pleural effusion.
5. Pregnant or breastfeeding women.
6. Patients planned for ECMO treatment.
7. Patients currently participating in or previously enrolled in other clinical studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Impact of low tidal volume vs airway pressure release ventilation on Dynamic relative regional lung strain（DRRS） | Maximum 4 hours

SECONDARY OUTCOMES:
mechanical power（MP） | Maximum 4 hours
platform pressure | Maximum 4 hours
mean airway pressure | Maximum 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Protti A, Cressoni M, Santini A, Langer T, Mietto C, Febres D, Chierichetti M, Coppola S, Conte G, Gatti S, Leopardi O, Masson S, Lombardi L, Lazzerini M, Rampoldi E, Cadringher P, Gattinoni L. Lung stress and strain during mechanical ventilation: any safe threshold? Am J Respir Crit Care Med. 2011 May 15;183(10):1354-62. doi: 10.1164/rccm.201010-1757OC. Epub 2011 Feb 4. PMID 21297069